CLINICAL TRIAL: NCT06309745
Title: THERApy De-escalation for TESTicular Cancer
Acronym: THERATEST
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: THERATEST
Record Dates: First submitted 2023-09-08; First posted 2024-03-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Seminoma
MeSH Terms: conditions — Seminoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RPLND cohort: Patients with seminoma who are negative/low for tumour markers and unifocal ipsilateral Stage IIA or <3cm IIB will be assessed for rRPLND. Patients who are eligible for rRPLND will undergo surgery followed by adjuvant treatment or surveillance as determined by their clinical teams based on post-operative histology as per SOC. Patients who are not deemed eligible for or decline rRPLND, will be offered either BEP/EP chemotherapy or radiotherapy with or without neoadjuvant Carboplatin AUC7 and will continue to be followed in the study.
  Interventions: Procedure: retroperitoneal lymph node dissection
- Carboplatin AUC10 cohort: Patients with stage II seminoma will be offered Carboplatin AUC10. Those deemed ineligible for Carboplatin AUC10 or who decline this treatment option will be offered either BEP/EP chemotherapy or radiotherapy and will continue to be followed in the study.
  Interventions: Drug: Carboplatin AUC10

INTERVENTIONS:
Procedure: retroperitoneal lymph node dissection — retroperitoneal lymph node dissection
  Groups: RPLND cohort
Drug: Carboplatin AUC10 — Carboplatin AUC10
  Groups: Carboplatin AUC10 cohort

SUMMARY:
THERATEST is looking to collect data from 30 patients actively receiving de-escalation treatments or other standard of care treatments in two UK hospitals. THERATEST is a feasibility study to determine whether patients are willing to be recruited, the impact of de-escalation treatments on patients' cancers and quality of life, whether we should proceed with these treatments in a larger study, and if so how the study should be conducted. A feasibility study prepares the ground for a larger study and improves the chances of the subsequent study producing valuable evidence, and helps to avoid wasting precious resources on larger trials that are unlikely to be informative. We hope that information from THERATEST will bridge the current knowledge gap and allow clinicians to design bigger trials to actively compare the different treatment strategies.

DETAILED DESCRIPTION:
THERATEST is an observational cohort study of patients receiving SOC treatments (combination chemotherapy or radiotherapy) or de-escalated treatments (primary rRPLND or Carboplatin AUC10) treatments for stage II seminoma.

Potential patients will be identified and invited to join the THERATEST study. Patients will be allocated to the following cohorts based on whether the relevant mode of treatment is adopted as an institutional SOC in their respective institution:

A. rRPLND cohort: Patients with seminoma who are negative/low for tumour markers and unifocal ipsilateral Stage IIA or <3cm IIB will be assessed for rRPLND. Patients who are eligible for rRPLND will undergo surgery followed by adjuvant treatment or surveillance as determined by their clinical teams based on post-operative histology as per SOC. Patients who are not deemed eligible for or decline rRPLND, will be offered either BEP/EP chemotherapy or radiotherapy with or without neoadjuvant Carboplatin AUC7 and will continue to be followed in the study.

B. Carboplatin AUC10 cohort: Patients with stage II seminoma will be offered Carboplatin AUC10. Those deemed ineligible for Carboplatin AUC10 or who decline this treatment option will be offered either BEP/EP chemotherapy or radiotherapy and will continue to be followed in the study.

Chemotherapy treatment strategies and adjuvant treatments are left to the shared decision-making between treating clinician and patient and follow institutional SOC. In both cohorts patients will be followed up for 2 years after treatment completion or until death or withdrawal of consent, whichever is the earliest. Beyond the study period, patients will be follow up as per institutional SOC protocols as part of prospective institutional audits.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

1. Willing and able to provide written informed consent.
2. Male.
3. Age ≥ 16 years.
4. Histologically confirmed seminoma (biopsy/orchidectomy)
5. Clinical stage II (standard of care cross-sectional imaging).
6. Ability to comply with the protocol, including but not limited to, completion of the patient-reported outcome questionnaires.

rRPLND cohort specific inclusion criteria

Participants must meet the following additional inclusion criteria to register for the rRPLND cohort:

1. Stage IIA and <3cm IIB with unifocal ipsilateral lymph node within rRPLND template.
2. Negative or mildly elevated serum tumour markers, defined as:

   1. AFP (alpha-fetoprotein) <10ng/ml and non-rising on serial testing
   2. BhCG (human chorionic gonadotropin) <50mg/ml
   3. LDH (lactate dehydrogenase) <1.5x upper limit normal
3. Fit for surgery, defined as meeting all of the following criteria:

   1. Body mass index (BMI) <34
   2. Charlson comorbidity index ≤3
   3. ECOG Performance status 0-1
   4. No significant cardio-pulmonary disease, or other uncontrolled intercurrent illness that would limit fitness for surgery in the opinion of the investigator
   5. No previous open intra-abdominal surgery

Carboplatin AUC10 cohort specific inclusion criteria

Participants must meet the following additional inclusion criteria to register for the Carboplatin AUC10 group:

1. Serum tumour markers, defined by IGCCCG "good risk" criteria:

   1. AFP <10ng/ml
   2. any BhCG
   3. LDH <2.5x ULN
2. Glomerular filtration rate by EDTA clearance over 25 ml/min (a measured creatinine clearance using Cockcroft and Gault would be allowed if unable to perform EDTA clearance).
3. ECOG Performance status 0-2.
4. Patients must be sterile or agree to use adequate contraception during the period of therapy.

Exclusion Criteria:

1. Raised AFP > 10ng/ml that does not fall to <10ng/ml following orchidectomy
2. Previous chemotherapy or radiotherapy for the disease under study.
3. Previous or concurrent malignancy other than testicular cancer, unless treated with curative intent and with no known active disease present for ≥2 years before enrolment and felt to be at low risk for recurrence by the treating physician (for example: non-melanoma skin cancer or lentigo maligna; breast ductal carcinoma in situ; prostatic intraepithelial neoplasia; urothelial papillary non-invasive carcinoma or urothelial carcinoma in situ).
4. Any condition that, in the opinion of the investigator, would interfere with evaluation of study intervention or interpretation of patient safety or study results such as medical comorbidities impacting on QoL or medical conditions or other disorders that would affect adherence to study requirements

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A. rRPLND cohort: Patients with seminoma who are negative/low for tumour markers and unifocal ipsilateral Stage IIA or <3cm IIB will be assessed for rRPLND. Patients who are eligible for rRPLND will undergo surgery followed by adjuvant treatment or surveillance as determined by their clinical teams based on post-operative histology as per SOC. Patients who are not deemed eligible for or decline rRPLND, will be offered either BEP/EP chemotherapy or radiotherapy with or without neoadjuvant Carboplatin AUC7 and will continue to be followed in the study.
  B. Carboplatin AUC10 cohort: Patients with stage II seminoma will be offered Carboplatin AUC10. Those deemed ineligible for Carboplatin AUC10 or who decline this treatment option will be offered either BEP/EP chemotherapy or radiotherapy and will continue to be followed in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-10-02 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
FEASIBILITY of recruitment and retention | through study completion, an average of 3 year
  To demonstrate feasibility of recruitment and retention (number of participants recruited per month and retained annually). Completion of recruitment of 30 patients into the THERATEST study, and measurement of overall patient retention within the trial until the 2-year follow-up visit.

SECONDARY OUTCOMES:
QUALITY OF LIFE assessed by difference in HRQOL scores | through study completion, an average of 3 year
  To determine differences in Health-related QOL (HRQOL) before and after treatment(s). Change in domain scale scores/single item scores in European Organisation for Research and Treatment of Cancer (EORTC) QLQ-TC26 and EORTC QLQ-C30, measured from baseline until the 2-year follow-up visit.
QUALITY OF LIFE assessed by difference in differences in sexual drive, function, and overall satisfaction | through study completion, an average of 3 year
  To determine differences in sexual drive, function, and overall satisfaction before and after treatment(s). Change in domain scale scores/single item scores in Brief Male Sexual Function Inventory (BMSFI), QLQ-TC26, and supplementary questions on retrograde ejaculation. Measured from baseline until the 2-year follow-up visit.
Progression free SURVIVAL | through study completion, an average of 3 year
  • To determine progression-free survival (PFS) and overall survival (OS) rates ensuring these fall in line with standard of care treatments outcomes (>95%). PFS rate at 2 years, defined as the proportion of patients who did not experience disease progression or death from any cause during the 2-year follow-up period.
OVERALL SURVIVAL | through study completion, an average of 3 year
  • To determine progression-free survival (PFS) and overall survival (OS) rates ensuring these fall in line with standard of care treatments outcomes (>95%). OS rate at 2 years, defined as the proportion of patients who did not experience death from any cause during the 2-year follow-up period.
SAFETY and complication of all treatments | through study completion, an average of 3 year
  • To assess the safety and complications of all treatments. Incidence, nature and severity of adverse events with severity determined according to CTCAE v5.0 collected from consent until 6 weeks post-surgery or chemotherapy.
  Surgical complications will be assessed by the Clavien-Dindo scoring system, and analysing details of surgical complications, blood transfusion, ITU admission and dialysis rates from patient records up to 6 months post-rRPLND.

CONTACTS AND LOCATIONS:
Overall Officials: Prabhakar Rajan, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts and London Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No